CLINICAL TRIAL: NCT07107243
Title: Speaking Valves With Transtracheal End-expiratory Pressure Measurement Predicts Upper Airway Patency in Prolonged Tracheostomy Patients: A Multicenter, Prospective Study
Brief Title: SV With TTPEE Measurement Predicts Upper Airway Patency in Prolonged Tracheostomy Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Hongying Jiang, MD, Sponsor-Investigator, Capital Medical University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2025-hxkfzx-dzx-001
Record Dates: First submitted 2025-07-22; First posted 2025-08-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-07

CONDITIONS: Tracheostomy
Keywords: transtracheal end-expiratory pressure; speaking valve; upper airway; prolonged tracheostomized patients
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Intervention Model Description: All patients received the speaking valve combined with the transtracheal end-expiratory pressure measurement protocol and bronchoscopy.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- True positive group (Experimental): Upper airway non-patency is defined as positive; otherwise, it is negative. The true positive group is defined as those for whom both the results of the speaking valve (SV) with the transtracheal end-expiratory pressure (TTPEE) measurement protocol and the bronchoscopy are positive.
  Interventions: Diagnostic Test: Speaking valve combined with airway pressure; Diagnostic Test: Bronchoscopy
- False positive group (Experimental): Upper airway non-patency is defined as positive; otherwise, it is negative. The false positive group is defined as the group in which the result of the speaking valve (SV) with the transtracheal end-expiratory pressure (TTPEE) measurement protocol is positive, and the result of the bronchoscopy is negative.
  Interventions: Diagnostic Test: Speaking valve combined with airway pressure; Diagnostic Test: Bronchoscopy
- True negative group (Experimental): Upper airway non-patency is defined as positive; otherwise, it is negative. The true negative group is defined as those for whom both the results of the speaking valve (SV) with the transtracheal end-expiratory pressure (TTPEE) measurement protocol and the bronchoscopy are negative.
  Interventions: Diagnostic Test: Speaking valve combined with airway pressure; Diagnostic Test: Bronchoscopy
- False negative group (Experimental): Upper airway non-patency is defined as positive; otherwise, it is negative. The false negative group is defined as the group in which the result of the speaking valve (SV) with the transtracheal end-expiratory pressure (TTPEE) measurement protocol is negative, and the result of the bronchoscopy is positive.
  Interventions: Diagnostic Test: Speaking valve combined with airway pressure; Diagnostic Test: Bronchoscopy

INTERVENTIONS:
Diagnostic Test: Speaking valve combined with airway pressure — All patients wore speaking valves for 30 minutes, during which the transtracheal end-expiratory pressure was measured to assess the patency of the upper airway.
Diagnostic Test: Bronchoscopy — The same examiner performed bronchoscopy on all patients to assess upper airway patency.

SUMMARY:
The aim of this study is to evaluate the feasibility of predicting upper airway patency in patients with prolonged tracheostomy using a non-invasive method combining speaking valve (SV) and transtracheal end-expiratory pressure (TTPEE) through a multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* Weaned from ventilator more than 48 hours
* No any organ failure
* No sepsis
* Stable heart rate and blood pressure
* Lung infection under control
* PCO2<60mmHg
* Patient and family sign informed consent form

Exclusion Criteria:

* Serious dysfunction of vital organs
* Inability to tolerate cuff deflation
* Laryngopharyngeal trauma
* Known severe upper airway obstruction before referrer to our department
* Endoscopy(bronchoscopy or laryngoscopy) has been performed and the condition of the upper airway has known

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of SV with transtracheal end-expiratory pressure measurement in predicting upper airway patency | The patients started using the SV with the TTPEE measurement on the day of enrollment. After that, bronchoscopy should be performed within 48 hours.
  Patients enrolled in the study will undergo both SV with transtracheal end-expiratory pressure measurement and bronchoscopy. Upper airway non-patency will be defined as positive. Using the results of bronchoscopy as the gold standard, the sensitivity and specificity of SV with transtracheal end-expiratory pressure measurement will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Hongying Jiang, MD, Study Chair — Beijing Rehabilitation Hospital of Capital Medical University
Locations (5):
- China (5):
  - Hunan Rehabilitation Hospital, Hunan, Hunan
  - Jiangbin Hospital of Guangxi Zhuang Autonomous Region, Guangxi, Jiangbin
  - Beijing Rehabilitation Hospital of Capital Medical University, Beijing, Shijingshan
  - YanBian University Hospital, Jilin, Yanbian
  - Zhengzhou Central Hospital Affiliated to Zhengzhou University, Henan, Zhengzhou

IPD SHARING:
Plan to Share IPD: No